CLINICAL TRIAL: NCT02764489
Title: A Phase 3b/4, Prospective, Multicenter, Open-label, Randomized, Crossover Study of Tolerability and Safety of FEIBA Reconstituted in Regular or 50% Reduced Volume and of Faster Infusion Rates in Patients With Hemophilia A or B With Inhibitors
Brief Title: FEIBA Reconstitution Volume Reduction and Faster Infusion Study (FEIBA STAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 091501; 2015-005781-39 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-05-06 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Hemophilia A or B With Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1:FEIBA 85±15 U/kg at Regular Volume Then 50% Reduced Volume at 2 U/kg/min Rate or Vice Versa (Experimental): Participants who were eligible were randomized to receive: 3 infusions (infusions 1, 2 and 3) of factor eight inhibitor bypassing activity (FEIBA) 85 ± 15 U/kg, reconstituted in regular volume sterile water for injection (SWFI) followed by 3 infusions (infusions 4, 5 and 6) of FEIBA 85 ± 15 U/kg reconstituted in 50% reduced volume SWFI (Sequence A) or: 3 infusions (infusions 1, 2 and 3) of FEIBA 85 ± 15 U/kg, reconstituted in 50% reduced volume SWFI, followed by 3 infusions of FEIBA 85 ± 15 U/kg, reconstituted in regular volume SWFI (Sequence B). All infusions in Part 1 were given at the standard infusion rate of 2 U/kg/min.
  Interventions: Biological: FEIBA
- Part 2:FEIBA 85±15U/kg 50% Reduced Volume at 4U/kg/min Rate Then at 10U/kg/min Rate (Experimental): Participants who completed Part 1, received FEIBA 85 ± 15 U/kg, reconstituted in 50% reduced volume SWFI at an increased rate of 4 U/kg/min for infusions 7, 8, and 9, followed by FEIBA 85 ± 15 U/kg, reconstituted in 50% reduced volume SWFI at an increased rate of 10 U/kg/min for infusions 10, 11, and 12.
  Interventions: Biological: FEIBA

INTERVENTIONS:
Biological: FEIBA — Anti-inhibitor Coagulant Complex Nanofiltered (activated prothrombin complex concentrate [APCC]), FEIBA NF.
  Other Names: FEIBA NF.; AICC; anti-inhibitor coagulant complex; Anti-inhibitor Coagulant Complex Nanofiltered (activated prothrombin complex concentrate [APCC]); APCC; Activated prothrombin complex concentrate

SUMMARY:
The purpose of this study is to:

* 1. To evaluate the tolerability and safety of infusing reduced volume Factor Eight Inhibitor Bypassing Activity (FEIBA) at the standard infusion rate of 2 U/kg/min
* 2. To evaluate the tolerability and safety of infusing reduced volume FEIBA at increased rates of 4 and 10 U/kg/min, in comparison to the standard rate of 2 U/kg/min at the regular volume

DETAILED DESCRIPTION:
15 JUN 2020: The temporary enrollment stop of new patients into this study due to the COVID-19 pandemic has been lifted in one or more countries/sites, and the study is now again enrolling new patients. However, some countries/sites may still have paused the enrollment of new patients due to the pandemic.

23 APRIL 2020: Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to (> or =) 18 to less than or equal to (< or =) 65 years old at the time of screening.
2. Hemophilia A or B of any severity, with a documented > or = 3 months history of inhibitors (> or = 0.6 Bethesda units [BU]) requiring the use of bypassing agents (FEIBA or rFVIIa) prior to screening. Inhibitor level will be tested at screening if no documented history is available.
3. Hepatitis C virus (HCV) negative, either by antibody testing or polymerase chain reaction (PCR); or HCV positive with stable liver disease.
4. Human immune deficiency virus (HIV) negative; or HIV positive with stable disease and CD4 count > or = 200 cells per cubic millimetre (cell/mm3) at screening.
5. Adequate venous access.
6. Willing and able to comply with the requirements of the protocol.
7. If a female of childbearing potential, must have a negative blood pregnancy test and agrees to employ adequate birth control measures for the duration of the study, such as: a. Abstain from sexual intercourse, b. Use a reliable method of contraception (contraception such as an intrauterine device, barrier method [e.g., diaphragm or sponge; female condom not permitted] with spermicide, oral contraceptive, injectable progesterone, sub dermal implant), and have their male partner use a condom
8. If female of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria:

   1. Postmenopausal, defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with follicle-stimulating hormone levels within the laboratory-defined postmenopausal range or postmenopausal with amenorrhea for at least 24 months and on hormonal replacement therapy.
   2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, bilateral tubal ligation (with no subsequent pregnancy at least 1 year from bilateral tubal ligation), or bilateral salpingectomy.

Exclusion criteria:

1. Known hypersensitivity to FEIBA or any of its components.
2. Advanced liver disease (e.g., liver biopsy confirmed diagnosis of cirrhosis, portal vein hypertension, ascites, prothrombin time [PT] 5 seconds above upper limit of normal).
3. Planned elective surgery during participation in this study (excluding minor procedures that will not need preventative bleeding treatments, such as exchanges of peripherally inserted central catheters).
4. Platelet count less than (<) 100,000/ microliter (μL).
5. Taking Emicizumab (Hemlibra) for bleed prevention.
6. Clinical or laboratory evidence of disseminated intravascular coagulation based on medical history.
7. Prior history or evidence of thromboembolic event: acute myocardial infarction, deep vein thrombosis, pulmonary embolism, etc.
8. Diagnosis of advanced atherosclerosis, malignancy, and/or other diseases that may increase the participant's risk of thromboembolic complications.
9. Participant is taking any immunomodulating drug (e.g., corticosteroid agents at a dose equivalent to hydrocortisone greater than (>) 10 milligram per day (mg/day), or α-interferon) within 30 days prior to enrollment except anti-retroviral chemotherapy.
10. Herbal supplements that contain anti-platelet activity.
11. Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
12. Participant is a family member or employee of the investigator.
13. Clinically significant medical, psychiatric or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (3):
- University Hospital Center Zagreb, Zagreb, Croatia
- PHI Institute for Transfusion Medicine of Macedonia, Skopje, North Macedonia
- MV Sklifosovskyi Poltava Hematology, Poltava, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc34db2bf003ab459c3

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in Thailand, Malaysia, Algeria, Croatia, India, Poland, Turkey, and Ukraine from 12 February 2019 to 27 December 2021. Participants with a diagnosis of Congenital Hemophilia A were enrolled.
Pre-assignment Details: Participants received factor eight inhibitor bypassing activity (FEIBA) reconstituted in regular volume and FEIBA reconstituted in 50% reduced volume in a crossover fashion for Part 1 and FEIBA reconstituted in 50% reduced volume at escalated infusion rates for Part 2. Participants who completed Part 1 entered Part 2 of the study. A total of 45 participants were enrolled in the study out of which 33 participants received the study treatment.
Groups:
- Part 1: Sequence A-FEIBA 85±15U/kg in Regular Volume, Then FEIBA 85± 15U/kg in 50% Reduced Volume: Participants were first randomized to receive 3 infusions of FEIBA 85 ± 15 U/kg, IV reconstituted in regular volume SWFI at the standard rate of 2 U/kg/min, every 48 hours. Participants then received 3 infusions of FEIBA 85 ± 15 U/kg, IV reconstituted in 50% reduced volume SWFI, at the standard rate of 2 U/kg/min, every 48 hours.
- Part 1: Sequence B-FEIBA 85±15 U/kg in 50% Reduced Volume, Then FEIBA 85±15 U/kg in Regular Volume: Participants were first randomized to receive 3 infusions of FEIBA 85 ± 15 U/kg, IV reconstituted in 50% reduced volume SWFI, at the standard rate of 2 U/kg/min, every 48 hours. Participants then received 3 infusions of FEIBA 85 ± 15 U/kg, IV reconstituted in regular volume SWFI at the standard rate of 2 U/kg/min, every 48 hours.
Period: Part 1: Day 1 up to Day 16
Arm/Group | Part 1: Sequence A-FEIBA 85±15U/kg in Regular Volume, Then FEIBA 85± 15U/kg in 50% Reduced Volume | Part 1: Sequence B-FEIBA 85±15 U/kg in 50% Reduced Volume, Then FEIBA 85±15 U/kg in Regular Volume
Started | 17 | 16
Completed | 14 | 16
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Part 2: Day 19 up to Day 41
Arm/Group | Part 1: Sequence A-FEIBA 85±15U/kg in Regular Volume, Then FEIBA 85± 15U/kg in 50% Reduced Volume | Part 1: Sequence B-FEIBA 85±15 U/kg in 50% Reduced Volume, Then FEIBA 85±15 U/kg in Regular Volume
Started (Participants who completed Part 1 of the study entered Part 2 of the study:) | 14 | 16
Part 2: FEIBA 85±15U/kg 50% Reduced Volume at 4U/kg/Min Rate (Participants who completed Part 1 of the study received up to 3 infusions of FEIBA 85 ± 15 U/kg IV reconstituted in 50% reduced volume SWFI at an increased infusion rate of 4 U/kg/min, every 48 hours (infusions 7, 8, and 9).) | 14 | 16
Part 2: FEIBA 85±15U/kg 50% Reduced Volume at 10U/kg/Min Rate (Participants who completed Part 1 of the study and received up to 3 infusions (infusions 7, 8, and 9) at the rate of 4 U/kg/min in Part 2 received up to 3 infusions (10, 11, and 12) of FEIBA 85 ± 15 U/kg IV reconstituted in 50% reduced volume SWFI at an increased infusion rate of 10 U/kg/min, every 48 hours.) | 12 | 16
Completed | 12 | 16
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Groups:
- Part 1 + Part 2: Overall FEIBA Treatment: Part 1:
  Participants who were eligible were randomized to receive: 3 infusions (infusions 1, 2 and 3) of FEIBA 85 ± 15 U/kg, reconstituted in regular volume SWFI followed by 3 infusions (infusions 4, 5 and 6) of FEIBA 85 ± 15 U/kg reconstituted in 50% reduced volume SWFI (Sequence A) or: 3 infusions (infusions 1, 2 and 3) of FEIBA 85 ± 15 U/kg, reconstituted in 50% reduced volume SWFI, followed by 3 infusions of FEIBA 85 ± 15 U/kg, reconstituted in regular volume SWFI (Sequence B).
  All infusions in Part 1 were given at the standard infusion rate of 2 U/kg/min.
  Part 2:
  Participants who completed Part 1, received FEIBA 85 ± 15 U/kg, reconstituted in 50% reduced volume SWFI at an increased rate of 4 U/kg/min for infusions 7, 8, and 9, followed by FEIBA 85 ± 15 U/kg, reconstituted in 50% reduced volume SWFI at an increased rate of 10 U/kg/min for infusions 10, 11, and 12.
Arm/Group | Part 1 + Part 2: Overall FEIBA Treatment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Measure: Count of Participants; unit: Participants
Groups:
- Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate: Participants were randomized to receive 3 infusions of FEIBA 85 ± 15 U/kg, IV reconstituted in regular volume SWFI at the standard rate of 2 U/kg/min, every 48 hours (Participants in Sequence A: infusions 1, 2, and 3 and Participants in Sequence B: infusions 4, 5 and 6).
- Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate: Participants were randomized to receive 3 infusions of FEIBA 85 ± 15 U/kg, IV reconstituted in 50% reduced volume SWFI, at the standard rate of 2 U/kg/min, every 48 hours (Participants in Sequence A: infusions 4, 5, and 6 and Participants in Sequence B: infusions 1, 2 and 3).
- Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate: Participants who completed Part 1 of the study received up to 3 infusions of FEIBA 85 ± 15 U/kg IV reconstituted in 50% reduced volume SWFI at an increased rate of 4 U/kg/min, every 48 hours (infusions 7, 8, and 9).
- Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate: Participants who completed Part 1 of the study and received up to 3 infusions (infusions 7, 8, and 9) at the rate of 4 U/kg/min in Part 2 received up to 3 infusions (10, 11, and 12) of FEIBA 85 ± 15 U/kg IV reconstituted in 50% reduced volume SWFI at an increased infusion rate of 10 U/kg/min, every 48 hours.
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 8 | 7 | 1 | 4

2. Primary Outcome: Number of Participants With Any Hypersensitivity Reaction
Description: Number of participants with AEs particular to allergic-type hypersensitivity reactions were assessed. Clinical manifestations of hypersensitivity reactions included, but was not limited to skin rash, pruritus (itching), urticaria (hives), angioedema (for example, swelling of the lips and/or tongue) and anaphylactic reaction.
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 3 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Any Thromboembolic Event
Description: Participants with adverse events related to thromboembolic event were reported. Clinical manifestations of thromboembolic events included, but was not limited to myocardial infarction, deep vein thrombosis, pulmonary embolism, stroke and transitory ischemic attack.
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Any Infusion Site Reaction
Description: Infusion sites were monitored for pain, tenderness, erythema, and swelling. Infusion site evaluations were made by clinical staff or by the participant or caregiver.
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 2 | 1 | 0 | 0

5. Primary Outcome: Number of Participants With AEs Leading to Study Discontinuation
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 2 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Vital Signs Considered as AEs
Description: Number of participants with vital signs considered as AEs were assessed. Vital signs included body temperature (degree Celsius or degrees Fahrenheit [°C or °F]), respiratory rate (breaths/min), pulse rate (beats/min), and systolic and diastolic blood pressure (millimeter of mercury [mmHg]).
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Laboratory Assessments Considered as AEs
Description: Number of participants with Laboratory Assessments considered as AEs were assessed. Laboratory assessments included hematology, clinical chemistry, coagulation testing, serological testing, pregnancy testing, cluster differentiation 4 (CD4).
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Population: SAS included all participants who received at least one dose of IP (i.e., FEIBA). Participants were counted more than once in the arm groups. Participants counted in Part 1 regular volume and in Part 1 reduced volume were the same.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
Number analyzed (Participants) | 33 | 30 | 30 | 28
Participants | 2 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 7 days after the end of infusion (up to Day 41)
Description: At each visit investigator documented occurrence of adverse events(untoward medical occurrence in participant administered IP that does not necessarily have a causal relationship with treatment). SAS=participants receiving at least one dose of IP(FEIBA).
Arm/Group | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/33 | 1/30 | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 2/33 | 5/30 | 0/30 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate (N=33) | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate (N=30) | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate (N=30) | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate (N=28)
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:FEIBA 85 ± 15 U/kg Regular Volume at 2 U/kg/Min Rate (N=33) | Part 1:FEIBA 85±15 U/kg 50% Reduced Volume at 2 U/kg/Min Rate (N=30) | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 4 U/kg/Min Rate (N=30) | Part 2:FEIBA 85±15 U/kg 50% Reduced Volume at 10 U/kg/Min Rate (N=28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2
Headache (Nervous system disorders) | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT02764489/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02764489/SAP_001.pdf